CLINICAL TRIAL: NCT04133883
Title: A Study to Investigate if the Use of a Systematic Joint Examination (Ultrasound/Functional/Physical) Has an Impact on the Physician's Haemophilia Treatment Management Decision in Patients With Haemophilia
Brief Title: Impact on French Physician's Haemophilia Treatment Management Decision Based on Systematic Joint Examination
Acronym: A-MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Sobi.HAEM8-001
Record Dates: First submitted 2019-10-18; First posted 2019-10-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hemophilia A
Keywords: joint health
MeSH Terms: conditions — Hemophilia A | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Haemophilia A patients (Other): Treated on-demand or prophylaxis with any Factor VIII (FVIII) product, plasma derived or recombinant (conventional or extended-half life) FVIII, according to routine clinical practice.
  Interventions: Procedure: Ultrasound, Haemophilia Joint Health Score

INTERVENTIONS:
Procedure: Ultrasound, Haemophilia Joint Health Score — Systematic joint examinations of ankles, knees and elbows

SUMMARY:
This low interventional study aims to describe if and how the haemophilia treatment management decisions are impacted by a systematic joint examination (ultrasound, functional, physical) in patients with haemophilia A in France.

DETAILED DESCRIPTION:
The study will assess the behavior of the physicians with regards to haemophilia management decisions, and if systematic joint examination have an impact on their decisions. The main objective is to evaluate if the use of HEAD-US and Haemophilia Joint Health Score (HJHS) have an impact on these decisions. The study is classified as a low-interventional study due to mandated systematically assessment (HEAD-US, HJHS) on patients which may not be part of routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-40 years
* Haemophilia A patients treated with plasma-derived factor VIII (pdFVIII) or recombinant (conventional or extended half-life) factor VIII (rFVIII)
* At least one joint bleeding episode prior to inclusion
* Signed informed consent

Exclusion Criteria:

* Enrolment in another concurrent clinical interventional study, or intake of an Investigational Medicinal Product, within three months prior to inclusion in the study
* Presence of factor VIII antibodies (inhibitors) (≥0.60 Bethesda Unit [BU]/mL) at the latest available inhibitor test
* Joint surgery over the past year prior to inclusion in one of the following joints; left knee, right knee, left elbow, right elbow, left ankle and right ankle
* More than one joint replacement

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Changes in haemophilia management based on systematic joint examinations of ankles, knees and elbows with HJHS and HEAD-US | 12 months
  Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Elena Santagostino, Study Director — Swedish Orphan Biovitrum
Locations (20):
- France (20):
  - Swedish Orphan Biovitrum Research site, Angers
  - Swedish Orphan Biovitrum Research site, Bordeaux
  - Swedish Orphan Biovitrum Research site, Brest
  - Swedish Orphan Biovitrum Research site, Caen
  - Swedish Orphan Biovitrum Research site, Chambéry
  - Swedish Orphan Biovitrum Research site, Clermont-Ferrand
  - Swedish Orphan Biovitrum Research site, Dijon
  - Swedish Orphan Biovitrum Research site, Le Kremlin-Bicêtre
  - Swedish Orphan Biovitrum Research site, Lyon
  - Swedish Orphan Biovitrum Research site, Marseille
  - Swedish Orphan Biovitrum Research site, Montpellier
  - Swedish Orphan Biovitrum Research site, Nancy
  - Swedish Orphan Biovitrum Research site, Nantes
  - Swedish Orphan Biovitrum Reserach site, Paris
  - Swedish Orphan Biovitrum Research site, Poitiers
  - Swedish Orphan Biovitrum Research site, Reims
  - Swedish Orphan Biovitrum Research site, Rouen
  - Swedish Orphan Biovitrum Research site, Strasbourg
  - Swedish Orphan Biovitrum Research site, Toulouse
  - Swedish Orphan Biovitrum Research Site, Tours

IPD SHARING:
Plan to Share IPD: No